CLINICAL TRIAL: NCT02162797
Title: EFFECT OF ZINC SUPPLEMENTATION ON IMMUNE RECOVERY PROGRAM HIV PATIENTS WITH AN IPS MEDELLIN
Brief Title: Zinc Supplementation Effect on Immune Recovery in HIV Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CES University (Other)
Collaborators: IPS Fundación SIAM (Unknown)
Responsible Party: Principal Investigator, Heidy Contreras, Researcher, CES University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUPL002
Record Dates: First submitted 2014-05-29; First posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: HIV; AIDS; Immunological Deficiency; Inadequate Immune Recovery; Viral Replication
Keywords: HIV; AIDS; zinc; zinc supplement; immunological deficiency
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Seroconversion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo supplementation (Experimental): Intervention Group B: Patients who will orally receive a placebo for 3 months.
  Interventions: Dietary Supplement: Placebo supplementation
- zinc supplementation (Experimental): Intervention group A. Patients who will orally receive zinc for 3 months.
  Interventions: Dietary Supplement: Zinc supplementation

INTERVENTIONS:
Dietary Supplement: Zinc supplementation — Intervention group A: Patients who will orally receive zinc for 3 months.
  Other Names: Zinc Supplementation in Patients With HIV
  Arms: zinc supplementation
Dietary Supplement: Placebo supplementation — Intervention Group B: Patients who will orally receive a placebo for 3 months.
  Arms: Placebo supplementation

SUMMARY:
INTRODUCTION:

An adequate zinc supplementation is essential for a good immunological function. However, zinc deficiency is seen in more than 50% of adults infected with HIV. The safety and efficiency of zinc supplements in the progression of HIV is evaluated in the short-term.

HYPOTHESIS

Null hypothesis: Zinc supplementation does not improve the immunological recovery of HIV patients after three months of daily consumption.

Alternate hypothesis: Zinc supplementation improves the immunological recovery of HIV patients after three months of daily consumption

DETAILED DESCRIPTION:
GOAL:

To assess the effect of zinc supplementation in the natural history of HIV, emphasizing on the immunological recovery of patients in a health care provider program in Medellín in 2012.

METHODS:

A prospective, randomized, double-blind, controlled clinical trial will be conducted. The selected group will consist of male and female patients over 18 years of age, who comply with the inclusion criteria, with digital clinical history, in an HIV/AIDS program of a health care provider in Medellín. They will receive zinc supplements for 3 months. A comparison will be made between the immunological recovery among those patients taking the zinc supplement and those who are not. The CD4 lymphocytes value will be taken as an independent variable.

ELIGIBILITY:
Inclusion Criteria:

* Adults suffering from HIV/AIDS, over 18 years of age with first- and second-line antiretroviral therapy.
* Patients with two viral loads less than 40 copies/ml (viral supression) and a stable or inferior CD4 lymphocyte count.
* Patients with body mass index over 18.5 kg/m2.
* Patients without opportunistic diseases.

Exclusion Criteria:

* Pregnant women.
* Hospitalized patients with cognitive disability evaluated by a doctor.
* Patients who are unwilling to participate.
* Patients taking zinc supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Immunological Recovery | Three months
  Zinc supplementation is expected to enhance the immunological response of HIV+ patients. This can be demonstrated comparing the initial analysis with the final report (3 months later).
EFFECT OF ZINC SUPPLEMENTATION ON IMMUNE RECOVERY PROGRAM HIV PATIENTS | THREE MONTHS
  Compare the variation in levels of CD4 lymphocytes at baseline and three months after surgery (zinc or placebo) in each study patient.

CONTACTS AND LOCATIONS:
Overall Officials: Heidy Contreras, PhC., Principal Investigator — Researcher; Marcela Duque, MD., Principal Investigator — Researcher; Elsa Vásquez, Biologist, Principal Investigator — Researcher
Locations (1):
- Fundación SIAM, Medellín, Antioquia, Colombia